CLINICAL TRIAL: NCT05537935
Title: Low Dose Naltrexone (LDN) for the Treatment of Chronic Neuropathic Pain in Patients With Human Immunodeficiency Virus (HIV), a Prospective, Pragmatic, Open Label Clinical Trial
Brief Title: Low Dose Naltrexone for Pain in Patients With HIV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Anne Marie McKenzie-Brown, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004422
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus; Chronic Neuropathic Pain
Keywords: Low dose Naltrexone; Naltrexone; Pain
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Pain | interventions — Naltrexone; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Once a potential subject has been identified they may be contacted with information about the study in advance of their appointment in order to allow time for them to consider the study. A qualifying pain score will be confirmed with the subject prior to initiating consent. This may occur up to 30 days before the baseline, treatment visit, but inclusion/exclusion criteria will be re-confirmed prior to initiating study treatment. Patients may also be approached during a clinic visit.
  Should a patient decline participation in the treatment plan, they will be invited to participate in a control group. They will be invited to complete the PROMIS questionnaire every 4 weeks, and the NPRS pain assessment every week from Baseline through week 12. These participants will receive follow up phone calls to confirm completion of these assessments weekly and will not have any in-person visits.
- Low Dose Naloxone (LDN) (Experimental): Once a potential subject has been identified they may be contacted with information about the study in advance of their appointment in order to allow time for them to consider the study. A qualifying pain score will be confirmed with the subject prior to initiating consent. This may occur up to 30 days before the baseline, treatment visit, but inclusion/exclusion criteria will be re-confirmed prior to initiating study treatment. Patients may also be approached during a clinic visit.
  Participants will start with 3mg LDN orally administered daily for one week, with a planned increase to 4 mg/day beginning week two, if tolerated. They will be provided with a four-week supply of study medication. LDN will be given as a daytime dose.
  Interventions: Drug: Low Dose Naltrexone

INTERVENTIONS:
Drug: Low Dose Naltrexone — Participants will start with 3mg LDN orally administered daily for one week, with a planned increase to 4 mg/day beginning week two, if tolerated. They will be provided with a 4-week supply of study medication. The most common side effects are difficulty sleeping and vivid dreams, which are seen more frequently with nighttime dosing, so LDN will be given as a daytime dose.
  Other Names: Questionnaires
  Arms: Low Dose Naloxone (LDN)

SUMMARY:
The increased life expectancy of Patients Living With HIV/AIDS (PLWHA) has increased the need for therapies for chronic conditions, such as chronic pain. Pain in the HIV population is often refractory and ends up being treated with chronic opioids, which are associated with adverse effects, including hyperalgesia, constipation, and risk of overdose. Naltrexone is an opioid antagonist used in the treatment of alcohol and opioid use disorders. Low Dose Naltrexone (LDN), naltrexone at a much lower dose, is thought to be an immune modulator and has been associated with an increased CD4 count in PLWHA. Repurposing this medication is relatively inexpensive and has the potential to expand access to treatment for a painful condition experienced in PLWHA. While there are many case reports on the efficacy of LDN in symptom reduction, there are only a small number of clinical trials that specifically examine pain and symptom relief.

This study will include patients who are not completely virologically controlled and will monitor the CD4 counts drawn as a part of routine care. If the CD4 count improves with LDN and with reduced symptoms, this could be a significant improvement in HIV therapy for symptom control. There have been studies showing cytokine reduction in fibromyalgia patients but they did not investigate the correlation with cytokines and pain relief. This study involves repurposing a drug used for substance use disorder to a medication with the potential to treat pain and improve symptoms for PLWHA.

DETAILED DESCRIPTION:
More than one million people in the United States live with HIV. In 2018, Black/African Americans made up 42% of the new HIV diagnoses, while Hispanic persons accounted for 27%. Black/African Americans and Hispanics with an HIV diagnosis receive less care for treatment and maintenance of HIV than their Caucasian counterparts and are thus less likely to have adequate suppression of the virus. Many people living with HIV/AIDS have untreated chronic pain, which negatively affects their quality of life. Neuropathic (nerve) pain, including painful HIV neuropathy, is notoriously difficult to treat. Opioids (narcotics) are often used to treat chronic pain in patients, with inconsistent results. We now know that opioids for chronic pain are more consistently known for a multitude of side effects than effective long-term pain relief. Lesser-known side effects of chronic opioids include suppressing, or dampening, the immune system, making opioids particularly undesirable as a chronic therapy for pain in the HIV patient population. Other therapies for neuropathic pain have undesirable side effects. Naltrexone is FDA-approved for addiction and is not used to treat a medical disease. Low-dose naltrexone (LDN) is an off-label use of naltrexone with some evidence that it may help chronic pain, such as fibromyalgia and some types of neuropathic (nerve) pain. LDN is a much lower dose of naltrexone. It has to be compounded to 1/10 of the usual dose to be repurposed to treat pain. In this study, 40 adult patients with HIV will take low-dose naltrexone for 12 weeks to treat neuropathic pain. We will measure pain scores and markers of inflammation while they are taking LDN. Naltrexone repurposed as LDN has the potential to greatly enhance the quality of life of HIV patients. This is particularly meaningful given the healthcare disparities often associated with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75, male and female
* HIV infection with a viral load of < 1000 copies/ml for the past six months. (That is the viral load below which, according to the 2018 American College of Obstetricians and Gynecologists (ACOG) Committee Opinion, there is not thought to be a significant risk of HIV transmission from the mother to the fetus with vaginal delivery. This was thought to be a reasonable cut-off for inclusion in this study.)
* Diagnosis of neuropathic pain (pain that is associated with a lesion or disease involving the somatosensory nervous system, e.g. painful neuropathy, radicular pain, complex regional pain syndrome, nerve-related pain following spine surgery, etc.) using the neuropathic pain screening tool, painDETECT17, as part of the neuropathic pain screen.
* Pain score > 4/10 on average on the NPRS lasting > 3 months (chronic pain)
* Capable of informed consent and willing to comply with the study requirements
* Fluent English-speaking

Exclusion Criteria:

* Allergy to naltrexone (not applicable to the control group)
* Current use of any opioids, up to 10 days before the start of the study (not applicable to the control group)
* Pregnant women
* Nursing mothers and women of childbearing potential not using contraception known to be highly effective (not applicable for the control group). Highly effective contraception methods include a combination of any two of the following during the 12-week study period:

  1. Use of oral, injected, or implanted hormonal methods of contraception or;
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  3. Barrier methods of contraception; condom or occlusive cap (diaphragm or cervical /vault caps) with spermicidal foam/gel/film/cream/vaginal suppository;
  4. Total abstinence;
  5. Male/female sterilization.
* Bipolar disorder, schizophrenia, poorly controlled anxiety or depression
* Diagnosis of liver disease, e.g. cirrhosis
* Current diagnosis of either chronic kidney disease or acute kidney injury and/or a GFR <45 at baseline
* Acute viral hepatitis A, B, C
* Patients who self-report as having tested positive for COVID-19 or have been diagnosed with another viral illness within the past ten days.
* Patients with a known or suspected diagnosis of long-term COVID
* Active drug or alcohol use disorder
* People who may require opioid therapy during the duration of the study, e.g. upcoming surgery
* Transportation issues interfering with return study visits (NA for the control group)
* Adults unable to consent
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Numerical Pain Score | Study weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10,11 and 12
  The study team will give participants a link to the online PROMIS questionnaire that includes a numerical pain rating scale (NPRS) to complete using an iPad or computer and will verbally ask questions to establish baseline information required for the study. If they have no computer access, they will be given a hard copy of the PROMIS questionnaire and NPRS to complete for future visits.
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
  Changes in pain scores, measured on the numerical pain score (NPS) on the Pain Intensity section of the PROMIS-29 Profile v2.0. This will be measured weekly during the 12-week study period.

SECONDARY OUTCOMES:
Changes in PROMIS pain Score | Study weeks 0, week 4, week 8 and week 12
  The study team will give participants the PROMIS questionnaire to complete using an iPad or computer, or a paper form, and will verbally ask questions to establish baseline information required for the study. If they have no computer access, they will be given a hard copy of the PROMIS questionnaire to complete for future visits.
  Changes in the overall score of the PROMIS-29 Profile v2.0 questionnaire collected at baseline, 4, 8, and 12 weeks will be assessed.
  The participants' answers to PROMIS-29 are scored from 1-5. The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score. PROMIS assessments use an Item Response Theory (IRT) based score called "Expected A Posteriori" or EAP scores, which are then transformed onto a final T-score metric. The scores are mapped so that the values follow a normal distribution with a population mean T-score of 50 and a standard deviation of 10.
Changes in Average pain Score | Study weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10,11 and 12
  The study team will give participants a link to the online PROMIS questionnaire that includes a numerical pain rating scale (NPRS) to complete using an iPad or computer and will verbally ask questions to establish baseline information required for the study. If they have no computer access, they will be given a hard copy of the PROMIS questionnaire and NPRS to complete for future visits.
  The study team will compare the average weekly pain scores of the study group with the control group.
Changes in IL-1 levels | Study week 0 and week 12
  Blood will be drawn by phlebotomy services according to institutional practice. Samples for will be sent to the Emory Medical Laboratory at EUH or Emory University Hospital Midtown (EUHM) for processing and analysis.
  Serum cytokines values will be measured at the 12-week visit and will be compared to baseline visit values.
Changes in IL-18 levels | Study week 0 and week 12
  Blood will be drawn by phlebotomy services according to institutional practice. Samples for will be sent to the Emory Medical Laboratory at EUH or Emory University Hospital Midtown (EUHM) for processing and analysis.
  Serum cytokines values will be measured at the 12-week visit and will be compared to baseline visit values.
Changes in Met-Enkephalin Levels | Study week 0 and week 12
  Blood will be drawn and collected by phlebotomy services according to institutional practices into 2 purple top tubes (EDTA, 10 ml) at the baseline and 12-week visits. These samples will be sent to the Emory Research Hemostasis and Coagulation Core Laboratory (ERHCCL) Changes in Met-Enkephalin levels at the 12-week visit compared to baseline visit levels.
Changes in endorphin levels | Study week 0 and week 12
  Blood will be drawn and collected by phlebotomy services according to institutional practices into 2 purple top tubes (EDTA, 10 ml) at the baseline and 12-week visits. These samples will be sent to the Emory Research Hemostasis and Coagulation Core Laboratory (ERHCCL) Changes in endorphin levels at the 12-week visit compared to baseline visit levels.
Changes in CD4 counts | Study week 0 and week 12
  Blood will be drawn and collected by phlebotomy services according to institutional practices into 2 purple top tubes (EDTA, 10 ml) at the baseline and 12-week visits. These samples will be sent to the Emory Research Hemostasis and Coagulation Core Laboratory (ERHCCL) Changes in CD4 counts levels at the 12-week visit compared to baseline visit levels.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M McKenzie-Brown, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Midtown Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal, to achieve aims of the approved proposal. ? Proposals may be directed to amckenz@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are available 5 years at a 3rd party website